CLINICAL TRIAL: NCT05002738
Title: Validation of 24-hour Trough Concentration as a Surrogate for Intensive Pharmacokinetic Measurements for a Combined Oral Contraceptive Pill Containing Desogestrel
Brief Title: Desogestrel-containing COCP Pharmacokinetic Validation Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 21-3936
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Contraception
MeSH Terms: interventions — Desogestrel; Ethinyl Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Overall Cohort (Experimental): Combined oral contraceptive pill containing 0.15mg desogestrel and 0.03mg ethinyl estradiol for 21 days
  Interventions: Drug: Desogestrel and Ethinyl Estradiol Tablets

INTERVENTIONS:
Drug: Desogestrel and Ethinyl Estradiol Tablets — Combined oral contraceptive pill

SUMMARY:
This study aims to validate prior pharmacokinetic research with combined oral contraceptive pill users that supports utilizing a 24-hour trough concentration as an accurate proxy for the intensive pharmacokinetic parameter of area under the curve (gold standard pharmacokinetics). The original pharmacokinetic studies were performed with a levonorgestrel-containing oral contraceptive pill and we aim to duplicate those findings with a desogestrel-containing oral contraceptive pill.

DETAILED DESCRIPTION:
Enrolled participants will be started on a standard pack of desogestrel-containing oral contraceptive pills and undergo an intensive pharmacokinetic study visit on day 21 of the pill pack. This will entail 11 serial blood draws and a final blood draw the next day at 24 hours post-pill intake to measure and calculate a pharmacokinetic area under the curve for both the estrogen and progestin components of the pill. We will then correlate the 24-hour trough measurement to the area under the curve measures to determine the correlation of these measurements.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females aged 18-45 years
* Body-mass index ≥18.5kg/m2
* Willing to abstain from medications and supplements known to induce/inhibit CYP3A4 during the study
* Normal blood pressure measurement at screening (systolic <140mmHg, diastolic <90mmHg)
* Negative urine pregnancy test at screening

Exclusion Criteria:

* Currently taking any known CYP3A4 inducers/inhibitors
* Medical conditions that affect liver function (e.g. hepatitis, cirrhosis)
* Any contraindications to estrogen-containing contraception (based on any category 3 or 4 recommendations from the CDC MEC guidelines)
* Use of an injectable contraceptive method within the last 6 months or current use of an ENG contraceptive implant
* Childbirth within the last 6 months
* Known allergy or insensitivity to combined oral contraceptive pills

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lazorwitz A, Sheeder J. Validation of 24-hour trough concentration as a proxy for intensive pharmacokinetic measurements for a combined oral contraceptive pill containing desogestrel. Contraception. 2023 Oct;126:110093. doi: 10.1016/j.contraception.2023.110093. Epub 2023 Jun 16. PMID 37331464

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Overall Cohort
Started | 22
Completed | 20
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Overall Cohort
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 28.3 [18.8 to 41.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body-mass index [Median (Full Range); unit: kg/m^2] | 24.8 [18.8 to 41.6]

OUTCOME MEASURES:

1. Primary Outcome: Serum Etonogestrel Concentrations
Description: 12 serum measurements taken over the course of 24 hours Correlation coefficient calculated for area under the curve versus 24-hour trough measurement
Time Frame: 24 hours
Measure: Number (95% Confidence Interval); unit: correlation coefficient (r)
Arm/Group | Overall Cohort
Number analyzed (Participants) | 20
correlation coefficient (r) | 0.92 [0.80 to 0.97]

2. Primary Outcome: Serum Ethinyl Estradiol Concentrations
Description: 12 serum measurements taken over the course of 24 hours Correlation coefficient calculated for area under the curve to 24-hour trough measurements
Time Frame: 24 hours
Measure: Number (95% Confidence Interval); unit: correlation coefficient (r)
Arm/Group | Overall Cohort
Number analyzed (Participants) | 20
correlation coefficient (r) | 0.86 [0.67 to 0.94]

ADVERSE EVENTS:
Time Frame: 22 days
Arm/Group | Overall Cohort
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT05002738/Prot_SAP_000.pdf